CLINICAL TRIAL: NCT06978049
Title: Use of Lactic Acid Gel for Intravaginal Use, 7 Applicators x 5ml, Bayer to Reduce Post-episiotomy Discomfort
Acronym: LA30051990
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Andrew Hospital Constanta (Other)
Collaborators: Ovidius University of Constanta (Other)
Responsible Party: Principal Investigator, Brezeanu Dragos, Principal Investigator, Ovidius University of Constanta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD30051990; 7230/31.01.2023 (Registry Identifier: Saint Andrew Hospital Ethical Comitee Registry)
Record Dates: First submitted 2025-04-25; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Episiotomy; Wound Healing; Postpartum Period
Keywords: Episiotomy; Wound Healing; Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canesbalance Group (Experimental): Participants in this group received topical lactic acid gel (a commercial product from BAYER, Bucharest, Romania) applied once daily directly to the episiotomy site. Treatment began on day 7 postpartum and continued for seven consecutive days.
  Interventions: Drug: Topical Lactic Acid Gel (BAYER)
- No Intervention Group (No Intervention): Participants in this group received standard postpartum care without the addition of lactic acid gel or any other specific wound-healing treatments. Healing occurred spontaneously according to routine clinical practice.

INTERVENTIONS:
Drug: Topical Lactic Acid Gel (BAYER) — Lactic acid gel, applied topically once daily to the episiotomy site, starting on postpartum day 7 for a total of seven consecutive days. Commercial product: BAYER (Bucharest, Romania).
  Arms: Canesbalance Group

SUMMARY:
This prospective controlled study evaluates the efficacy of topical lactic acid gel in enhancing episiotomy wound healing and improving postpartum sexual quality of life.

DETAILED DESCRIPTION:
This prospective controlled clinical study aims to evaluate the efficacy of topical lactic acid gel in promoting the healing of episiotomy wounds and improving postpartum sexual quality of life.

The study was conducted at the County Clinical Emergency Hospital "Sf. Ap. Andrei" in Constanța, Romania, between February 1, 2023, and December 31, 2024, with ethical approvals obtained from both the Ethics Committee of Ovidius University of Constanța (No. 01/20.01.2023) and the Saint Andrew Hospital Ethics Committee (No. 7230/31.01.2023).

A total of 100 postpartum women aged 18 to 40 years, who underwent spontaneous vaginal delivery with mediolateral episiotomy at a gestational age of 38-40 weeks, were enrolled in the study after providing informed consent. Participants were sequentially assigned into two parallel groups:

Experimental Group (n = 50): Received topical lactic acid gel (commercially available formulation from BAYER, Bucharest, Romania) applied once daily directly to the episiotomy site, starting seven days postpartum, for a total duration of seven consecutive days.

Control Group (n = 50): Received standard postpartum care without additional topical treatments, allowing for spontaneous healing of the episiotomy wound.

The primary endpoint was the assessment of episiotomy wound healing quality at 40 days postpartum, determined via visual inspection and healing scoring. The secondary endpoint was the evaluation of postpartum sexual function, assessed using a validated 12-item sexual quality of life questionnaire specifically designed for postpartum women. The questionnaire addressed domains including sexual desire, orgasm frequency, sexual satisfaction, pain during intercourse (dyspareunia), vaginal dryness, emotional well-being during intercourse, and partner-related factors. Higher total scores reflected better sexual health and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Spontaneous vaginal delivery with mediolateral episiotomy at 38-40 weeks gestation
* No pre-existing wound healing disorders or infections
* Provided informed consent

Exclusion Criteria:

* Known hypersensitivity to lactic acid products
* Third- or fourth-degree perineal tears
* Gestational diabetes or immunosuppressive conditions
* Use of additional wound care treatments

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only postpartum women aged 18 to 40 years who have undergone spontaneous vaginal delivery with mediolateral episiotomy are eligible for inclusion in this study. Male participants are not eligible, as the study specifically investigates female perineal wound healing and postpartum sexual quality of life.
Enrollment: 100 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Episiotomy Wound Healing Score at 40 Days Postpartum | 40 days postpartum
  Evaluation of the quality of episiotomy wound healing, assessed through visual inspection and clinical scoring at 40 days postpartum. Higher scores reflect better wound healing. Healing assessment was performed by the clinical care team using a standardized evaluation system to ensure consistency across participants.

SECONDARY OUTCOMES:
Increase in Quality of Sexual Life | 40 days postpartum
  Healing outcomes and sexual quality of life wIll be assessed 40 days postpartum using a 12-item questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Andrew Hospital, Constanța, Constanța County, Romania

IPD SHARING:
Plan to Share IPD: No
The study involves sensitive personal health information, including sexual function and postpartum recovery data, which are subject to strict confidentiality and privacy regulations. Participant consent for public data sharing was not obtained, and sharing of individual-level data may pose risks to participant anonymity. Only aggregate results will be reported in publications.